CLINICAL TRIAL: NCT07028060
Title: The Detection of Lung Pathologies Among Dialysis Patients Using Novel Mobile-Phone Ultrasound - A Feasibility Pilot Study
Brief Title: Detection of Lung Pathologies Among Dialysis Patients Using Pulsenmore MC™ Device - Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseNmore (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0539-20-SOR
Record Dates: First submitted 2022-11-28; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hemodialysis Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic renal failure patients (Experimental): All patients diagnosed with End-stage renal disease (ESRD) and treated with chronic dialysis center at Soroka University Medical Center (SUMC)
  Interventions: Device: PulseNmore MC™

INTERVENTIONS:
Device: PulseNmore MC™ — novel mobile Self-scan ultrasound device, Pulsenmore MC™

SUMMARY:
PRIMARY OBJECTIVE: To measure success rate and identification of pathological lung B-lines, using novel mobile Self-scan ultrasound device (MC, by Pulsenmore), in chronic renal failure patients, pre and post dialysis.

SECONDARY OBJECTIVE: 1.To describe the difference in B-lines score (BLS), pre and post dialysis as measured by the new device.

2. Examine the degree of agreement in the BLS performed by the new mobile , MC device to the traditional POCUS device.

3. To describe the identification rate of lung atelectasis and pleural effusion by the study device compared to standard ultrasound machine STUDY DESIGN: A prospective, pilot, single-center study. INTERVENTION: Lung point of care ultrasound (POCUS) performed with a new ultrasound device, MC based on mobile phone among chronic renal failure patients pre and post dialysis. SAMPLE SIZE CONSIDERATIONS: As this is a feasibility study sample size was not calculated, we will perform convenience sample of 30 patients.

STUDY PROCEDURES: Lung point of care ultrasound (POCUS) performed with a new MC device on chronic renal failure patients pre and post dialysis.

The following data will be collected:

* Demographic factors: age, gender, ethnicity
* Medical history: medications, diabetes mellitus, hypertension, systemic diseases, Congestive Heart Failure (CHF), Chronic Obstructive Pulmonary Disease (COPD), height and weight
* Clinical data:

oDates of admission oTreatment: dialysis duration (years) oEssential: heart rate, blood pressure, saturation, weight. Dry weight, BMI. All before and after session

* US results- BLS detected from pictures collected by:

  o the new MC device o the traditional POCUS device
* Detection of lung atelectasis by o the new MC device o the traditional POCUS device
* Detection of pleural effusion by o the new MC device o the traditional POCUS device

OUTCOMES AND ANALYSES:

* Agreement rate between the study MC device and the gold standard ultrasound machine for primary and secondary objectives.
* Time of study in each machine.

DETAILED DESCRIPTION:
Background Patients with end-stage renal disease (ESRD) and heart failure (HF) have a high risk to suffer from pulmonary congestion (PC) (1,2). PC in HF and ESRD patients is a common cause of admission, mortality, and cardiac events )3-6(. Extravascular lung water (EVLW), which leads to PC, can be subclinical among normo-hydrated dialysis patients (1,7).

PC exact mechanism in ESRD is under debate )8( but occurs in a combination of two forces mechanism - changes in hydrostatic pressure due to HF and volume overload and increase in lung permeability with retention of uremic product and chronic inflammation (1,2,6,8). Chronic load of extracellular volume and increased LV filling pressure is mainly the cause of EVLW accumulation leading to clinical PC (1,2). Volume overload builds gradually during the interval between the dialysis treatments (6,7) and maybe asymptomatic (1,6). PC can also occur in ESRD patients, even with normal cardiac filling pressure or mild volume overload )8( and can be explained by volume redistribution (2). Untreated or suboptimal treated PC can cause respiratory distress. Volume overload is an independent risk factor for death and cardiovascular events in ESRD patients (2,9). Therefore, volume removal is crucial to prevent PC events (2). Dialysis reduces the severity of PC immediately )8(, and delay in treatment can increase the frequency and the severity of the events (8,9).

Lung ultrasound (LUS) is an effective, bedside, imaging tool for the detection and monitoring of PC (2,7-12). Alveolar interstitial syndrome, which can be caused by an increase of EVLW, is diagnosed by the detection of ultrasonographic B-lines in both lung zones (2,3,5,7,9,10). Lung ultrasound was found at least sensitive and effective as other traditional modalities to diagnose PC (1,4,5,8,10,13).

B-lines are hyperechoic reverberation, relatively simple to teach and conduct (3,8,11), which can be detected by LUS (5,8,14). Some studies quantified B-lines using the B-line score (BLS). The score is calculated by the number of lung zones that are dichotomously positive for B-lines (10,11). Furthermore, B-lines are an important prognostic factor for death, cardiovascular events, and readmission in ESRD and HF patients (2-4,10-12).

Changes in BLS seen during volume removal by dialysis treatment or diuresis (2,7-10) represents the dynamic changes in EVLW (7,9-11). Studies found a distinct real-time decrease in the number of B-line and BLS that correlated with the traditional examination for EVLW (2,9- 11,13). Data suggests that B-lines monitoring is used for the assessment of volume overload removal adequacy (2,4,10,11).

A tool that can help the patients to manage their disease better, by early, self- identification of evolving PC, can shorten time to definite treatment (2,9). This may lead to reduced hospitalization and improved patients' clinical outcome.

In the present study, the investigators sought to check the feasibility of a new mobile US probe device that connects to a mobile phone, on hemodialysis patients. The investigators will compare the results measured by the new device to the traditional US device.

Ultrasound is very potent in the identification of these lung pathologies. The investigators would like to identify the sensitivity and specificity of this device in the detection of these other lung pathologies.

5 Method: Prospective, single center, pilot study will be carried out at the SUMC, and Soroka Clinical Research Center (SCRC), will oversee and manage the study.

5.1 Working Hypothesis

1. The study device, a novel mobile phone-based ultrasound device, Pulsenmore MC can identify B lines in high sensitivity and specificity and can replace traditional bigger and more expensive ultrasound machines for this diagnosis.

   5.2 Objective 5.2.1 Primary Objective To measure success rate and identification of pathological lung B-lines, using novel mobile phone, Pulsenmore MC device, in chronic renal failure patients, pre and post dialysis.

   5.2.2 Secondary Objective
   * To describe the difference in B-lines score (BLS), pre and post dialysis as measured by the new device.
   * Examine the degree of agreement in the BLS performed by the new mobile Pulsenmore MC device to the traditional ultrasound device.

   5.4 The study population will be screened at SUMC nephrology ward before scheduled dialysis. Population will be enrolled according to the following inclusion and exclusion criteria.

   5.4.1 Inclusion Criteria • Patients diagnosed with End-stage renal disease (ESRD) and treated with chronic dialysis center at Soroka University Medical Center (SUMC)
   * Cognitive intact and can sign informed consent as decided by their treating nephrologist.
   * have smart phone and any social app- like WhatsApp- his or her main care giver 5.4.2 Exclusion Criteria
   * Morbid obese - BMI>35
   * History of lung resection or lung transplant. 5.4.3 Withdrawal Criteria All patients should be encouraged to remain in the study through both of the ultrasound test. However, if a patient decides to discontinue study participation, the reason for discontinuation must be recorded in the medical record and the Case Report Form (CRF).

   5.5 Enrollment 5.6 Patient Screening Screening will be performed at the dialysis center located in the nephrology. Interested patients will be asked to provide written consent prior to performing any study procedure.

   5.7 Study Procedures 5.7.1 Screening informed consent and Enrollment, training patient on the Pulsenmore MC device and then save the images from new mobile MC device and from the traditional POCUS device (Standard of care US equipment). After the enrollment of the first 10 patients, Additional 20 patients will be enrolled and receive the new ultrasound device, MC, that connects to the mobile phone. Till 24 hours before dialysis treatment, those patients will perform a self-examination at home using the demo or the video guided mode. . . The patients will receive instruction on how to use the device. The duration of the study, for these patients, will be up to three weeks (6-10 dialysis).

   At Screening and enrollment visit: The patient will be consented after examination with inclusion and exclusion criteria.

   Demographics, Medical History, Clinical data, device details, and vital signs data will be collected.

   The patient will be trained on Pulsenmore MC device. Patient will receive instructions how to use the new ultrasound device and when to self-scan himself.

   First dialysis treatment in the study can be performed on the same day of subject consent.

   Dialysis treatments (6-10):

   US images will be recorded and documented before and after the dialysis from 3 zones (and both sides - right and left) Two physicians will analyze the data from the Self-scan ultrasound device compared to the traditional ultrasound device.

   AE and CCMED will be reviewed.

   Phase I: In- clinic: dialysis unit, enrolment of max 10 patients receiving ES or MC for up to 3 weeks of use (6-10 dialysis sessions). Each patient will be weighed Before & after Dialysis

   Study procedure -Before Dialysis:

   • Physician training
   * Physician with Patient: watching the tutorials
   * Physician scanning the patient for B lines and lung pathologists using the Demo or the video guided mode MC - scanning both sides.
   * Patient scanning for B lines using the Pulsenmore MC Demo or the video guided mode - scanning both sides.
   * Later, on the same day, the patients will have an in-person clinic visit and will be scanned by a physician/technician for lung pathologies using the Standard of care US equipment. The scanned images, from demo or the video guided mode, will be uploaded to the cloud from the patient 's device and interpreted by 2 physicians.

   Study procedure - After Dialysis:
   * Physician scanning for B lines using MC
   * Physician scanning for B lines using the Standard of care US.

   Phase II: At Home: enrolment of 20 patients receiving MC for up to 3 weeks of use (6-10 dialysis).

   *A patient who participate in the first phase will also be able to participate in the second phase of the study. Each patient will be weighed Before & after Dialysis

   Study procedure -Before Dialysis:
   * Physician training in clinic using the Demo or the video guided mode.
   * Physician with Patient: watching the tutorials or Practice scan.
   * Patient scanning for B lines using MC in Demo or video guided mode, scanning both sides. This procedure will be performed at home, till 24 hours before dialysis treatment.
   * Later, on the same day, the patients will have an in-person clinic visit and will be scanned by a physician/technician for lung pathologies using the Standard of care US equipment.

   Study procedure - After Dialysis:

   • Physician scanning for B lines using MC

   • After using the MC, Physician scanning for B lines using the Standard of care US.

   • The in-clinic scan serves as Ground truth (GT).

   • At the end of phase 1 or 2, the images from the Demo scan or the video guided mode, will be uploaded to the cloud from the patient 's device and interpreted by 2 physicians.

   5.8 Study Duration: the investigators expect that enrollment to the study will be for a period of 10 months.

   5.9 Data to Capture 5.9.1 Required Data All required data for this study will be collected via electronic case report forms (eCRF).

   5.9.2 Data Collection The final set of CRFs is designed to accommodate the specific features of the trial design. Modification of CRFs will only be made if deemed necessary by Soroka CRC. The CRFs will be filled out manually by the study personal and or will be collected through the computer services database.

   The following data will be collected:

   • Demographic factors: age, gender, ethnicity

   • Medical history: medications, diabetes mellitus, hypertension, systemic diseases, Congestive Heart Failure (CHF), Chronic Obstructive Pulmonary Disease (COPD), height and weight

   • Clinical data:

   -Dates of admission

   -Treatment: dialysis duration (years)

   -Essential: heart rate, blood pressure, saturation, weight in Kg, Before and after session, Dry weight and BMI.

   US results - from pictures collected from New mobile Pulsenmore MC and standard device (Traditional US POCUS) before and after the dialysis from 3 zones (and both sides right and left)

   -BLS, pleural effusion and lung atelectasis from each device and each zone Each patient will receive the same code for both devices' records for blinded comparison that All the analysis of BLS will be decided by an independent blinded reviewer.

6. Statistical Considerations and Analysis Plan 6.1 Statistical Analyses Data will be expressed as mean SD, median, and interquartile range, or as percent and frequency, as appropriate.

All statistical tests and/or confidence intervals, as appropriate, will be performed at α=0.05 (2-sided). All p-values reported will be rounded to three decimal places.

6.2 Sample Size Considerations We will analyze data of all relevant patients who meet all the inclusion criteria and none of the exclusion criteria. This feasibility research we will perform on 30 different patients.

6.3 Primary Endpoints Comparison between the devices in the b-lines test. Number of b lines, more than 2, more than 5, confluent 6.4 Secondary Analyses and Endpoints

Secondary end point:

6.4.1. Comparison of lung pathologies of both sides, right and left, between Pulsenmore MC and Standard of care US devices for pleural effusion, atelectasis, and consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients diagnosed with End-stage renal disease (ESRD) and treated with chronic dialysis center at Soroka University Medical Center (SUMC)
* Cognitive intact and can sign informed consent as decided by their treating nephrologist.
* have smart phone and any social app- like WhatsApp- his or her main care giver

Exclusion Criteria:

* Morbid obese - BMI>35
* History of lung resection or lung transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
To measure success rate and identification of pathological lung B-lines, using novel mobile phone, Pulsenmore MC device, in chronic renal failure patients, pre and post dialysis. | 10 months
  To measure success rate and identification of pathological lung B-lines, using novel mobile phone, Pulsenmore MC device, in chronic renal failure patients, pre and post dialysis.

SECONDARY OUTCOMES:
To describe the difference in B-lines score (BLS), pre and post dialysis as measured by the new device, Pulsenmore MC | 10 months
  To describe the difference in B-lines score (BLS), pre and post dialysis as measured by the new device, Pulsenmore MC
Examine the degree of agreement in the BLS performed by the new mobile Pulsenmore MC device to the traditional ultrasound device. | 10 months
  Examine the degree of agreement in the BLS performed by the new mobile Pulsenmore MC device to the traditional ultrasound device.
To describe the identification rate of lung atelectasis and pleural effusion by the study | 10 months
  To describe the identification rate of lung atelectasis and pleural effusion by the study

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency care unit, Beersheba, Israel

REFERENCES:
- [Background] Mallamaci F, Benedetto FA, Tripepi R, Rastelli S, Castellino P, Tripepi G, Picano E, Zoccali C. Detection of pulmonary congestion by chest ultrasound in dialysis patients. JACC Cardiovasc Imaging. 2010 Jun;3(6):586-94. doi: 10.1016/j.jcmg.2010.02.005. PMID 20541714
- [Background] Saad MM, Kamal J, Moussaly E, Karam B, Mansour W, Gobran E, Abbasi SH, Mahgoub A, Singh P, Hardy R, Das D, Brown C, Kapoor M, Demissie S, Kleiner MJ, El Charabaty E, El Sayegh SE. Relevance of B-Lines on Lung Ultrasound in Volume Overload and Pulmonary Congestion: Clinical Correlations and Outcomes in Patients on Hemodialysis. Cardiorenal Med. 2018;8(2):83-91. doi: 10.1159/000476000. Epub 2017 Nov 29. PMID 29617006
- [Background] Cogliati C, Casazza G, Ceriani E, Torzillo D, Furlotti S, Bossi I, Vago T, Costantino G, Montano N. Lung ultrasound and short-term prognosis in heart failure patients. Int J Cardiol. 2016 Sep 1;218:104-108. doi: 10.1016/j.ijcard.2016.05.010. Epub 2016 May 13. PMID 27232920
- [Background] Covic A, Siriopol D, Voroneanu L. Use of Lung Ultrasound for the Assessment of Volume Status in CKD. Am J Kidney Dis. 2018 Mar;71(3):412-422. doi: 10.1053/j.ajkd.2017.10.009. Epub 2017 Dec 21. PMID 29274919
- [Background] Gargani L, Sicari R, Raciti M, Serasini L, Passera M, Torino C, Letachowicz K, Ekart R, Fliser D, Covic A, Balafa O, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Shavit L, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Kraemer TD, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Onofriescu M, Zarzoulas F, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. Efficacy of a remote web-based lung ultrasound training for nephrologists and cardiologists: a LUST trial sub-project. Nephrol Dial Transplant. 2016 Dec;31(12):1982-1988. doi: 10.1093/ndt/gfw329. Epub 2016 Sep 26. PMID 27672089
- [Background] Torino C, Gargani L, Sicari R, Letachowicz K, Ekart R, Fliser D, Covic A, Siamopoulos K, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Gueler F, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Siriopol D, Balafa O, Shavit L, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. The Agreement between Auscultation and Lung Ultrasound in Hemodialysis Patients: The LUST Study. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2005-2011. doi: 10.2215/CJN.03890416. Epub 2016 Sep 22. PMID 27660305
- [Background] Liang XK, Li LJ, Wang XH, Wang XX, Wang YD, Xu ZF. Role of Lung Ultrasound in Adjusting Ultrafiltration Volume in Hemodialysis Patients. Ultrasound Med Biol. 2019 Mar;45(3):732-740. doi: 10.1016/j.ultrasmedbio.2018.10.025. Epub 2018 Dec 14. PMID 30558830
- [Background] Sherman RA. Crackles and Comets: Lung Ultrasound to Detect Pulmonary Congestion in Patients on Dialysis is Coming of Age. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):1924-1926. doi: 10.2215/CJN.09140816. Epub 2016 Sep 22. No abstract available. PMID 27660304
- [Background] Miglioranza MH, Gargani L, Sant'Anna RT, Rover MM, Martins VM, Mantovani A, Weber C, Moraes MA, Feldman CJ, Kalil RA, Sicari R, Picano E, Leiria TL. Lung ultrasound for the evaluation of pulmonary congestion in outpatients: a comparison with clinical assessment, natriuretic peptides, and echocardiography. JACC Cardiovasc Imaging. 2013 Nov;6(11):1141-51. doi: 10.1016/j.jcmg.2013.08.004. Epub 2013 Oct 2. PMID 24094830
- [Background] Ross DW, Abbasi MM, Jhaveri KD, Sachdeva M, Miller I, Barnett R, Narasimhan M, Mayo P, Merzkani M, Mathew AT. Lung ultrasonography in end-stage renal disease: moving from evidence to practice-a narrative review. Clin Kidney J. 2018 Apr;11(2):172-178. doi: 10.1093/ckj/sfx107. Epub 2017 Sep 28. PMID 29644056
- [Background] Martindale JL. Resolution of sonographic B-lines as a measure of pulmonary decongestion in acute heart failure. Am J Emerg Med. 2016 Jun;34(6):1129-32. doi: 10.1016/j.ajem.2016.03.043. Epub 2016 Mar 19. PMID 27061502
- [Background] Miglioranza MH, Picano E, Badano LP, Sant'Anna R, Rover M, Zaffaroni F, Sicari R, Kalil RK, Leiria TL, Gargani L. Pulmonary congestion evaluated by lung ultrasound predicts decompensation in heart failure outpatients. Int J Cardiol. 2017 Aug 1;240:271-278. doi: 10.1016/j.ijcard.2017.02.150. PMID 28606680
- [Background] Annamalai I, Balasubramaniam S, Fernando ME, Srinivasaprasad ND, Suren S, Thirumalvalavan K, Veerakumar AM. Volume Assessment in Hemodialysis: A Comparison of Present Methods in Clinical Practice with Sonographic Lung Comets. Indian J Nephrol. 2019 Mar-Apr;29(2):102-110. doi: 10.4103/ijn.IJN_78_18. PMID 30983750